CLINICAL TRIAL: NCT02563340
Title: Efficacy and Safety of Bone Marrow-derived Mesenchymal Stem Cells (BM-MSCs) on Chronic Antibody-mediated Rejection (cAMR) After Kidney Transplantation: A Multi-center Perspective Study
Brief Title: Effect of BM-MSCs on Chronic AMR After Kidney Transplantation
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Collaborators: Second Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Changxi Wang, Director of Organ Transplant Center, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MSC-KTx-cAMR-150926
Record Dates: First submitted 2015-09-26; First posted 2015-09-30 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2015-09

CONDITIONS: Kidney Transplantation
Keywords: kidney transplantation; antibody-mediated rejection; mesenchymal stem cell therapy; donor specific antibody; acute rejection
MeSH Terms: interventions — Desensitization, Psychologic; Immunoglobulins, Intravenous; Rituximab; Bortezomib

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- MSCs group (Experimental): cAMR patients in this group receive additional intravenous allogeneic BM-MSCs (1*10^6/kg) every two weeks for four consecutive doses, besides current desensitization therapy including at least one of the following treatments: plasmapheresis (PP), intravenous immunoglobulin (IVIG), rituximab or Bortezomib.
  Interventions: Other: BM-MSCs; Other: Desensitization therapy (PP, IVIG, rituximab or Bortezomib)
- Control group (Active Comparator): cAMR patients in this group receive current desensitization therapy including at least one of the following treatments: plasmapheresis (PP), intravenous immunoglobulin (IVIG), rituximab or Bortezomib.
  Interventions: Other: Desensitization therapy (PP, IVIG, rituximab or Bortezomib)

INTERVENTIONS:
Other: BM-MSCs — BM-MSCs are from third-party healthy donors, and have no HLA alleles similar to renal allograft donors or reacting to positive anti-HLA antibodies in recipients.
  Other Names: allogeneic bone marrow-derived MSCs
  Arms: MSCs group
Other: Desensitization therapy (PP, IVIG, rituximab or Bortezomib) — At least one drug or treatment is applied as desensitization therapy to decrease DSA, reduce B cells or inhibit plasma cells, depending on individual condition.

SUMMARY:
This study is designed to investigate the efficacy and safety of allogeneic bone marrow-derived mesenchymal stem cells (BM-MSCs) on chronic antibody-mediated rejection (cAMR) after kidney transplantation. Chronic AMR is diagnosed according to Banff criteria 2013 based on renal graft biopsy and donor specific antibodies (DSA) examination. cAMR patients are assigned to MSCs group or control group. Patients in control group are prescribed to current desensitization therapy including at least one of the following treatments: plasmapheresis (PP), intravenous immunoglobulin (IVIG), rituximab or Bortezomib, depending on individual pathological and immunological features (eg. DSA type and titer) of each study subjects. Patients in MSCs group receive additional BM-MSCs therapy besides desensitization treatments as in control group. Allogeneic BM-MSCs (1*10^6/kg) are intravenously administered every two weeks for four consecutive doses. All cAMR patients are followed up for one year. Renal function, DSA level, pathological features, patient/graft survival, and severe adverse events are monitored during the follow-up period. Immunological features of patients in both groups are consecutively examined.

ELIGIBILITY:
Inclusion Criteria:

* kidney transplantation
* cAMR diagnosis is determined based on renal graft biopsy and DSA examination
* Patient is willing and capable of giving written informed consent for study participation and able to participate in the study for 12 months

Exclusion Criteria:

* Combined or multi-organ transplantation
* Women who are pregnant, intend to become pregnant in the next 1 years, breastfeeding, or have a positive pregnancy test on enrollment or prior to study medication administration
* Donors or recipients are known hepatitis C antibody-positive or polymerase chain reaction (PCR) positive for hepatitis C
* Donors or recipients are known hepatitis B surface antigen-positive or PCR positive for hepatitis B
* Donors or recipients are known human immunodeficiency virus (HIV) infection
* Patients with active infection
* Recipients with a history of substance abuse (drugs or alcohol) within the past 6 months, or psychotic disorders that are not capable with adequate study follow- up
* Patients with severe cardiovascular dysfunction
* WBC<3*10^9/L or RBC <5g/dL
* Highly allergic constitution or having severe history of allergies
* Patients with active peptic ulcer disease, chronic diarrhea, or gastrointestinal problem affect absorption
* Patients with a history of cancer within the last 5 years
* Prisoner or patients compulsorily detained (involuntarily incarcerated) for treatment or either a psychiatric or physical (e.g. infectious disease) illness
* Renal graft function deteriorates due to non-immunological complication, such as surgical issues or drug nephrotoxicity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-10 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Estimated glomerular filtration rate (eGFR) | 12 months
  eGFR at month 12 after enrollment

SECONDARY OUTCOMES:
Patient survival rate | 12 months
  patient survival rate at month 12 after enrollment
Graft survival rate | 12 months
  graft survival rate at month 12 after enrollment
Donor specific antibody (DSA) level | 12 months
  Change of DSA level up to 12 months after enrollment
Pathological manifestation | 12 months
  Change of pathological scores according to Banff 2013 criteria
Severe adverse events | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Changxi Wang, M.D., Ph.D, Study Chair — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Peng Y, Ke M, Xu L, Liu L, Chen X, Xia W, Li X, Chen Z, Ma J, Liao D, Li G, Fang J, Pan G, Xiang AP. Donor-derived mesenchymal stem cells combined with low-dose tacrolimus prevent acute rejection after renal transplantation: a clinical pilot study. Transplantation. 2013 Jan 15;95(1):161-8. doi: 10.1097/TP.0b013e3182754c53. PMID 23263506
- See also: Previous publication — http://www.ncbi.nlm.nih.gov/pubmed/23263506